CLINICAL TRIAL: NCT02011789
Title: A Pilot Study To Determine The Metabolism And Health Effects Of Citrus Limonoids in Hypercholesterolemic Human Subjects
Brief Title: Metabolism And Health Effects Of Citrus Limonoids in Hypercholesterolemic Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: The Beverage Institute for Health & Wellness (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FL45
Record Dates: First submitted 2013-12-04; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; inflammation; citrus limonoids
MeSH Terms: conditions — Hypercholesterolemia; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group1 (Experimental): Group 1 consumes Placebo beverage for 56 days followed by Citrus Limonoid Beverage for 56 days.
  Interventions: Dietary Supplement: Citrus Limonoid Beverage; Dietary Supplement: Placebo beverage
- Group 2 (Active Comparator): Group 2 consumes Citrus Limonoid Beverage for 56 days followed by Placebo beverages for 56 days
  Interventions: Dietary Supplement: Citrus Limonoid Beverage; Dietary Supplement: Placebo beverage

INTERVENTIONS:
Dietary Supplement: Citrus Limonoid Beverage — The limonoid containing beverage will be 12-oz buffered, sterile, orange flavored, artificially sweetened, containing 60 mg vitamin C, 11 mg riboflavin and 250 mg limonin glucoside.
Dietary Supplement: Placebo beverage — The placebo beverage will be 12-oz buffered, sterile, orange flavored, artificially sweetened, containing 60 mg vitamin C and 11 mg riboflavin.

SUMMARY:
Limonoids are compounds found in citrus juices, seeds and peel. Some research shows that they reduce blood cholesterol and also reduce the incidence of several forms of cancer. Although these compounds are part of the natural human diet, the dose required to provide health benefits and the risks associated with the intake of high doses by humans have not been studied. This study will examine metabolism, safety, lipid-lowering and anti-inflammatory effects of limonoids. The dose of limonoids in this study is equivalent to that found in six 8 oz glasses of orange juice per day. The investigators hypothesize that limonin glucoside supplementation will reduce total cholesterol, LDL cholesterol, ratio of LDL and HDL cholesterol, number of LDL particles, and serum markers of inflammation.

DETAILED DESCRIPTION:
This is a 127-day study with a cross-over design, divided into three metabolic periods (P1, P2, and P3). For the first 14 days (P1), all subjects will receive two placebo beverages and will be asked to consume one each with breakfast and dinner. Then in metabolic period 2 (P2), subjects will be randomly assigned to one of two groups (Group 1 and Group 2). For the next 56 days, Group 1 will continue to consume two placebo beverages per day, while Group 2 will consume two beverages containing limonoids (250 mg/beverage). During the final 56 days (P3), the beverages provided to Group 1 will contain limonoids, and beverages provided to Group 2 will be placebo. Both the placebo and limonoid beverages will be 12-oz buffered, sterile, orange flavored, artificially sweetened beverage, containing 60 mg vitamin C, 11 mg riboflavin and zero calories. Subjects are instructed that they must drink all the beverage provided each day. Beverages will contain a biomarker (riboflavin), and the biomarker is assayed in urine samples collected every 2 weeks at the beverage pickup appointments to monitor compliance. The subjects will be informed that they are being monitored for compliance. Limonin glucoside is obtained from citrus waste materials utilizing chromatographic methods that employ food grade approved media and solvents. The final pure limonin glucoside is fractionally crystallized from a concentrated water solution of a chromatographically purified extract. The crystalline material is separated from the mother liquor, dried and subjected to mass spectral and nuclear magnetic resonance assessment. The spectral data is compared to data acquired for a pure limonin glucoside standard to establish final purity which is better than 95%.

Blood samples (approximately 70 ml, less than five tablespoons) will be drawn after a 12 hour overnight fast on study days 1, 15, 71 and 127 by venipuncture. These blood samples will be used to determine serum limonoids, complete blood cell count (CBC), and comprehensive chemistry panel (CCP), serum lipids, markers of inflammation, lymphocyte and monocytes functions. In addition to the fasting blood draws on days 15 (Group 2) and day 71 (Group 1), repeated blood samples (5 ml each time, approximately one teaspoon) will be drawn at 2, 4, 6, 8, and 24 hr after taking two 12-oz limonoid beverages (total limonoids 500mg) to determine the absorption and metabolism of limonoids. The investigators note that the blood samples drawn 24-h after the limonoid intake will be on study day 16 for Group 2 and day 72 for Group 1. The total amount of blood drawn will be less than 500 ml (2 cups) in 127 days. A spot urine sample will be collected at the same visit as the fasting blood draws, and every two weeks at the beverage pickup appointments. Repeated blood draws at 0, 2, 4, 6, and 8 hr after the limonoid supplement will be accompanied by the collection of urine samples. No food will be allowed during the 8 hrs; water intake will be monitored and restricted to one liter. Subjects will be served two standardized meals during this time, each representing 35% of their daily caloric intake, one after the 0 hr blood draw and the other after the 8 hr blood draw.

Subjects will be instructed not to change their diets, exercise or lifestyle during the course of the study. They will also be instructed not to consume any citrus fruit/juice (orange, grape fruit) throughout the study. Three 24-hour dietary recalls will be collected by telephone during the last week of each metabolic period (P1, P2, P3). A standardized diet will be served for all three meals for each day prior to the blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Hypercholesterolemic, total blood cholesterol 200-300 mg/dL
* BMI 20-35 kg/m2
* normal Complete Blood Count
* normal serum transaminases, alkaline phosphatase, and creatinine
* normal thyroid function
* LDL cholesterol > 130 mg/dL
* Triglyceride < 300 mg/dL
* serum C-Reactive Protein 1.0-25 mg/L

Exclusion Criteria:

* current pregnancy or lactation
* smoking
* use of alcohol > 1 drink per day (1 oz distilled liquor, 3 oz wine, 12 oz beer)
* reported history of cardiovascular disease or chronic inflammatory diseases
* current users of oral contraceptives
* lipid-lowering, anti-inflammatory, anti-coagulant, or thyroid medications
* currently drinking more than 4 glasses per day of orange or grapefruit juice

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in plasma lipids | 1, 15, 71 and 127 days
  Plasma cholesterol, LDL-cholesterol, HDL-cholesterol, triglyceride (TG), and remnant chylomicron particle concentrations will be determined. Lipid particle sizing will be performed by using nuclear magnetic resonance (NMR) technology. Plasma concentrations of apoproteins A1, B, C-III, and E will be measured.

SECONDARY OUTCOMES:
Change in liver and renal function | 1, 15, 71 and 127 days
  Serum sodium, potassium, chloride, carbon dioxide, urea nitrogen, creatinine, glucose, calcium, protein, albumin, alkaline phosphatase, asparagine transaminase (AST), bilirubin, alanine transaminase (ALT), and lactate dehydrogenase (LDH) were performed at the Pathology Laboratory of the University of California Davis Medical Center to assess liver and renal function.

OTHER OUTCOMES:
Change in inflammatory markers | 1, 15, 71 and 127 days
  Plasma concentrations of c-reactive protein (CRP), tumor necrosis factor (TNF-alpha), interleukin-1 (IL-1beta) and interleukin-6 (IL-6) will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Darshan S Kelley, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (1):
- USDA Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- See also: United States Department of Agriculture, Western Human Nutrition Research Center — http://www.ars.usda.gov/main/site_main.htm?modecode=53-06-25-00